CLINICAL TRIAL: NCT04362800
Title: Functional Effects and Impact on Motor Neuronal Activity of Early and Intensive MOtrice (Hand and Arm Bimanual Intensive Therapy Including Lower Extremities: HABIT-ILE) Reeducation in Children With Pre-school Bilateral Cerebral Palsy: a Trial Multicentre Randomized Control With Medico-economic Evaluation
Brief Title: Functional Effects and Impact on Motor Neuronal Activity of Early and Intensive Motrice (Hand and Arm Bimanual Intensive Therapy Including Lower Extremities: HABIT-ILE) Reeducation in Children With Pre-school Bilateral Cerebral Palsy
Acronym: MOOV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MOOV (29BRC20.0046)
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy (CP); pre-school children with bilateral CP
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): 10 days of intensive and structured motor therapy, 5 hours a day = 50h
  Interventions: Other: MRI; Other: Electro-Encephalography-High Density; Other: 3D and EMG analysis; Other: care and classic activities
- Control (Placebo Comparator): 10 days of care and classic activities
  Interventions: Other: MRI; Other: Electro-Encephalography-High Density; Other: 3D and EMG analysis; Other: care and classic activities

INTERVENTIONS:
Other: MRI — MRI at baseline and J90
Other: Electro-Encephalography-High Density — Electro-Encephalography-High Density (children with unilateral PC only) at baseline and J90
Other: 3D and EMG analysis — 3D and EMG analysis at baseline and J90
Other: care and classic activities — physiotherapy and psychomotility. As needed weekly sessions of speech therapist or orthoptist and daily activities of the child.

SUMMARY:
One of the urgent priorities in the field of pediatric neuro-rehabilitation is the development of efficient early motor interventions for children with cerebral palsy (CP). Animal studies suggest that early intensive interventions are likely to have a significant impact on the organization of the brain and corticospinal tracts, reducing motor impairments and their medium and long-term consequences in children with cerebral palsy. Although most of the growth, development and cortical organization takes place in the time course of the first 2 years of life, most studies investigating the effectiveness of intensive rehabilitation and associated neurophysiological mechanisms have been conducted in school-aged children (> 6 years). In addition, the vast majority of these studies were conducted in children with unilateral CP, while the bilateral form of the pathology has the highest prevalence. It is therefore a priority to investigate the effectiveness of early interventions on the overall motor function of children with CP, especially in children with bilateral form of CP.

Hand and Arm Bimanual Intensive Therapy Including Lower Extremities (HABIT-ILE) makes it possible to apply the concepts of structured motor learning and intensive treatment to both the upper limbs and the lower limbs and demonstrated improvements at both levels in school-aged children with unilateral CP and bilateral and then at all three International Classification of Functioning and Disability levels. The principles and content of HABIT-ILE can be applied to pre-school children and this method is promising for early neuro-rehabilitation.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate the effect of 10 days (i.e. 50 hours) of early HABIT-ILE (HABIT-ILE) on the overall motor function of children aged 1 to 4 with bilateral cerebral palsy in comparison to 10 days (50h) of spontaneous overall motor activity including usual rehabilitation (control group).

ELIGIBILITY:
Inclusion Criteria:

* Child with bilateral cerebral palsy proven to be spastic or dyskinetic
* 1 to 4 years old inclusive (12 to 59 months) (age corrected if premature) able to follow instructions and to be able to carry out all the assessments, in accordance with his age
* Being matched to a child according to age, etiology of CP / classification of motor function (GMFCS)
* Signature of consent by the two holders of parental authority

Exclusion Criteria:

* Exceed 4 years and 11 months (59 months) during the internship evaluation period.
* Uncontrolled epilepsy.
* History of toxin injection or surgery in the 6 months preceding the study period or scheduled within 3 months (during the study period).
* Visual or cognitive deficit preventing the child from seeing the games and interacting
* Usual contraindications to magnetic resonance imaging (MRI) such as metal implants.

Ages: 12 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2021-09-17 (Actual); Study Completion 2021-09-17 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Measure (GMFM) | 1 hour
  Measures change in gross motor function over time in children with cerebral palsy. The score range from 0 to 100 as a percentage. 100 is the best outcome.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Les Capucins, Angers
  - Fondation ILDYS - Site de Ty Yann, Brest

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.